CLINICAL TRIAL: NCT00626080
Title: Effects of INsulin dEtemiR and Neutral protaminE Hagedorn (NPH) Insulin on BRain glucOse Metabolism: a Study in Persons With Type 1 Diabetes
Brief Title: Insulin Detemir Action in Cerebro
Acronym: INcEREBRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: M. Diamant, VU University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DC2007Det001; 2007-007255-13
Record Dates: First submitted 2008-02-19; First posted 2008-02-29 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Type 1 Diabetes
Keywords: Insulin; Detemir; Brain; Glucose metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Detemir; Insulin, Isophane; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin detemir — 100 IU/ml, QD, dose individually adjusted, to be used for a period of 12 weeks; in combination with insulin aspart TID
  Other Names: Insulin Levemir
Drug: Insulin NPH — 100 IU/ml, QD, dose individually adjusted, to be used for a period of 12 weeks; in combination with insulin aspart TID
  Other Names: Insulin Insulatard

SUMMARY:
The aim of this study is to test the hypothesis that subcutaneous administration of insulin detemir, as compared to insulin NPH, leads to a more pronounced effect on cerebral glucose metabolism and/or cerebral blood flow in brain regions associated with appetite regulation, to account for the reported difference in weight.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patients;
* Diabetes duration =/> 1 year;
* HbA1c ~ 7,5%;

Exclusion Criteria:

* Recent onset of DM;
* BMI < 18 OR > 35 kg/m2;
* T2DM;
* History of major heart/renal disease;
* Severe untreated proliferative retinopathy;
* History of recurrent severe hypoglycaemia;
* (History of) brain disorders;
* Alcohol abuse,(History of) drug abuse, benzodiazepines, selective beta-blockers, oral steroids, oral anticoagulants;
* Current psychiatric disease/treatment;
* (history of) eating disorders;
* History of severe head trauma accompanied by loss of consciousness;
* Any endocrine disease not well controlled for at least 3 months;
* Inability to undergo MRI;
* Visual acuity < 0.3;
* Known or suspected allergy to trial product or related products

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cerebral metabolic rate of glucose, in brain regions associated with appetite control, as determined by FDG-PET | After 12 weeks of treatment
Cerebral blood flow, in brain regions associated with appetite control, as determined by H2O-PET | After 12 weeks of treatment

SECONDARY OUTCOMES:
CSF insulin concentration | After 12 weeks of treatment
Activity in brain regions associated with appetite control, as determined by fMRI | After 12 weeks of treatment
Weight change | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Diamant, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] van Golen LW, Veltman DJ, IJzerman RG, Deijen JB, Heijboer AC, Barkhof F, Drent ML, Diamant M. Effects of insulin detemir and NPH insulin on body weight and appetite-regulating brain regions in human type 1 diabetes: a randomized controlled trial. PLoS One. 2014 Apr 16;9(4):e94483. doi: 10.1371/journal.pone.0094483. eCollection 2014. PMID 24739875
- [Derived] van Golen LW, IJzerman RG, Huisman MC, Hensbergen JF, Hoogma RP, Drent ML, Lammertsma AA, Diamant M. Cerebral blood flow and glucose metabolism in appetite-related brain regions in type 1 diabetic patients after treatment with insulin detemir and NPH insulin: a randomized controlled crossover trial. Diabetes Care. 2013 Dec;36(12):4050-6. doi: 10.2337/dc13-0093. Epub 2013 Oct 15. PMID 24130356
- [Derived] van Golen LW, Huisman MC, Ijzerman RG, Hoetjes NJ, Schwarte LA, Lammertsma AA, Diamant M. Cerebral blood flow and glucose metabolism measured with positron emission tomography are decreased in human type 1 diabetes. Diabetes. 2013 Aug;62(8):2898-904. doi: 10.2337/db12-1159. Epub 2013 Mar 25. PMID 23530004
- [Derived] Huisman MC, van Golen LW, Hoetjes NJ, Greuter HN, Schober P, Ijzerman RG, Diamant M, Lammertsma AA. Cerebral blood flow and glucose metabolism in healthy volunteers measured using a high-resolution PET scanner. EJNMMI Res. 2012 Nov 20;2(1):63. doi: 10.1186/2191-219X-2-63. PMID 23168248